CLINICAL TRIAL: NCT02812537
Title: Clinical and Social Trajectories of Children and Adolescents With Disruptive Behavior: Multidisciplinary Approach of Pediatric and Psychiatric Emergencies in the Rhône-Alpes Auvergne Region
Brief Title: Clinical and Social Trajectories of Children and Adolescents With Disruptive Behavior
Acronym: TRAJECTORIES
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL16_0136
Record Dates: First submitted 2016-06-13; First posted 2016-06-24 (Estimated); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Disruptive Behavior Disorder
Keywords: Trajectories; emergency room; conduct disorder; care management
MeSH Terms: conditions — Attention Deficit and Disruptive Behavior Disorders; Emergencies; Conduct Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients with conduct disorders: Girls and boys having less than 16 years old and admitted to emergency room for aggressiveness, violence, fugue or theft.
  Interventions: Other: patients with conduct disorders

INTERVENTIONS:
Other: patients with conduct disorders — interview with a specialist

SUMMARY:
Conduct disorders are defined as "repetitive and persistent pattern of behavior in which the basic rights of others or major age-appropriate norms are violated". So defined, these disorders are at the crossroads of psychiatry, social field and justice. Conduct disorder management is a public health issue and a societal question. Conduct disorders affect 5 to 9% of 15-year old boys.

Care management of children and adolescents admitted for disruptive behaviors in emergency rooms is an issue. No consensus or official recommendation exists. However, use of emergency care in this context is increasing in most western countries and it exposes to several risks (inappropriate use of hospitalizations, social rupture, ignorance of comorbidities and suicide risk). The Trajectories project is designed to describe children and adolescents with disruptive behaviors, their care management and to follow their life trajectory and psychiatric evolution after admission to emergency rooms. Better understanding this population will improve their medical and social care management, thereby giving professionals the right tools.

The main objective of this project is to implement a multidisciplinary and integrative research combining clinical considerations and social sciences to determine the "trajectory" of this population.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents less than 16 years old
* Children and adolescents admitted to emergency rooms for aggressiveness, violence, fugue or theft

Exclusion Criteria:

* Children and adolescents admitted to emergency rooms for a reason not directly link with aggressiveness, violence, fugue or theft
* Opposition to the subject or the family to participate to this research

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children and adolescents admitted to emergency rooms for conduct disorder (aggressiveness, violence, fugue or theft)
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-05-20 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Number of new admissions to emergency rooms for aggressiveness, violence, fugue or theft | 6 months
  Six months follow-up of these children and adolescents in their future trajectory after the first admission to emergency room for disruptive behavior

SECONDARY OUTCOMES:
Age of the children and adolescents admitted to emergency rooms for aggressiveness, violence, fugue or theft | Day 0
  mean age
Gender of the children and adolescents admitted to emergency rooms for aggressiveness, violence, fugue or theft | Day 0
Number of children and adolescents precisely diagnosed with " behavior/conduct disorder | Day 0
Number of hospitalization | Day 0
  following the admission
number of patients admitted to emergency rooms for aggressiveness | Day 0
number of patients admitted to emergency rooms for violence | Day 0
number of patients admitted to emergency rooms for fugue | Day 0
number of patients admitted to emergency rooms for theft | Day 0
number of suicide attempts | 24 months
number of patients with disruptive behavior recurrence | 24 months
evolution of the CBCL score | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Yannis Gansel, MD, Principal Investigator — Hospices Cicils de Lyon
Locations (1):
- Hospices Civils de Lyon, Bron, France

IPD SHARING:
Plan to Share IPD: No